CLINICAL TRIAL: NCT03387878
Title: A Multi-centre Clinical Investigation to Assess the Performance of GentleCath™ Glide Intermittent Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CC-925-17-U378
Record Dates: First submitted 2017-08-22; First posted 2018-01-02 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Comfort and Performance of Intermittent Catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Study (Other): This is a single arm study with no comparator
  Interventions: Device: Intermittent Catheter

INTERVENTIONS:
Device: Intermittent Catheter — Intermittent urinary catheter for bladder drainage

SUMMARY:
To evaluate the performance of GentleCath Glide™ Intermittent Catheters

ELIGIBILITY:
Inclusion Criteria:

* Subjects of 18 years old and above who require intermittent bladder drainage may be recruited into the study
* Subjects must be willing and able to provide written informed consent
* Subjects may be either inpatients or outpatients but must all be capable of completing a patient diary card to record study data
* Subjects must currently use intermittent catheters and have been using intermittent catheters for the last six months
* Patients who self-catheterise at least three times per day
* Able to attend final assessment visit at day 14

Exclusion Criteria

* Subjects who require intermittent catheterisation to administer irrigation or instillation.
* Subjects who are presently participating in another clinical trial.
* Subjects exhibiting any other medical condition which, according to the investigator, justifies the subject's exclusion from the study
* Subjects with known sensitivity to the device components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Performance/Ease of Use | 14 Days
  Performance and ease of use will be assessed by both the patient and Investigator. The data will be collected via a questionnaire. The responses will be on a 1 to 5 scale with 1 disagreeing with the statement and 5 agreeing with the statement
Ease of Removal | 14 Days
  Ease of removal will be assessed by both the patient and Investigator. The data will be collected via a questionnaire. The responses will be on a 1 to 5 scale with 1 disagreeing with the statement and 5 agreeing with the statement
Residue Acceptability | 14 Days
  Residue acceptability will be assessed by both the patient and Investigator. The data will be collected via a questionnaire. The responses will be on a 1 to 5 scale with 1 disagreeing with the statement and 5 agreeing with the statement

CONTACTS AND LOCATIONS:
Locations (1):
- Specjalistyczny Gabinet Lekarski, Rzeszów, Poland